CLINICAL TRIAL: NCT00635050
Title: Phase II Trial of Primary Systemic Therapy for Locally Advanced Breast Cancer Using Sequential Doxil, Paclitaxel, and Cyclophosphamide With Concurrent Avastin
Brief Title: Therapy for Locally Advanced Breast Cancer Using Doxil, Paclitaxel, and Cyclophosphamide With Avastin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Ortho Biotech, Inc. (Industry); Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, John Carpenter, MD, Professor, Medicine, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F070824009; UAB 0493 (Other: UAB)
Record Dates: First submitted 2008-03-06; First posted 2008-03-13 (Estimated); Results first posted 2016-06-15 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-06

CONDITIONS: Invasive Breast Cancer
Keywords: Breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — liposomal doxorubicin; Paclitaxel; Cyclophosphamide; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Doxil, Paclitaxel, Cyclophosphamide + Avastin (Experimental): Two stage phase II single arm trial to evaluate the pathologic complete response rate to sequential dose dense chemotherapy using Doxil 25 mg/M2 iv and Avastin 10 mg/kg iv every 2 weeks x 3, then paclitaxel 175 mg/M2 iv and Avastin 10 mg/kg iv every 2 weeks x 3, then cyclophosphamide 600 mg/M2 iv and Avastin 10 mg/kg iv every 2 weeks x 3, in patients with locally advanced invasive breast cancer.
  Interventions: Drug: Doxil, Paclitaxel, Cyclophosphamide, Avastin

INTERVENTIONS:
Drug: Doxil, Paclitaxel, Cyclophosphamide, Avastin — Regimen A: Doxil 25 mg/M2 iv and Avastin 10 mg/kg iv every 2 weeks x 3, then paclitaxel 175 mg/M2 i.v. and Avastin 10 mg/kg iv every 2 weeks x 3, then cyclophosphamide 600 mg/M2 i.v. and Avastin 10 mg/kg iv every 2 weeks x 3 . Patients who experience <pCR to primary chemotherapy will receive an additional year of Avastin 15 mg/kg iv every 3 weeks, beginning 6-8 weeks after operation.
  Regimen B: Doxil 30 mg/M2 iv and Avastin 10 mg/kg iv every 2 weeks x 3, then paclitaxel 175 mg/M2 i.v. and Avastin 10 mg/kg iv every 2 weeks x 3, then cyclophosphamide 600 mg/M2 i.v. and Avastin 10 mg/kg iv every 2 weeks x 3. Patients who experience <pCR to primary chemotherapy will receive an additional year of Avastin15 mg/kg iv every 3 weeks, beginning 6-8 weeks after operation.
  Other Names: Bevacizumab (Avastin)

SUMMARY:
This study will evaluate the rate of pathological complete response (pCR) to the sequential therapy of Doxil, paclitaxel, and cyclophosphamide with concurrent Avastin for patients with locally advanced invasive (T2,T3, Nany, M0) breast carcinoma. Also, the study will evaluate the clinical and subclinical cardiotoxic effect(s) of this regimen, assess how feasible and safe the study is. Survival without any progression of disease will also be calculated.

A regimen of chemotherapy will be given to replicate the high rate of pCR seen with conventional chemotherapy in patients with locally advanced breast cancer. Doxil will substitute the normally given doxorubicin. It is expected that the low effect or minimal effect of Doxil on cardiac function will minimize any additional risk of cardiotoxicity from Avastin. It is expected that clinical and subclinical rates of cardiotoxicity will be very low at the total doses to be given in this clinical trial.

DETAILED DESCRIPTION:
In this trial, an attempt will be made to replicate the high rate of pathological complete response seen after conventional chemotherapy in patients with locally advanced breast cancer, using a regimen in which Doxil is substituted for conventional doxorubicin. We expect that the low or minimal effect on cardiac function produced by Doxil will minimize any additional risk of cardiotoxicity from Avastin. We will also measure left ventricular ejection fractions before and after treatment to see if the substantial rate of subclinical cardiotoxicity reported by Swain et al 5 and Perez et al 7 can be avoided. The reported rates of cardiotoxicity after treatment with relatively high doses of Doxil are substantially lower than those of doxorubicin; few data are available to estimate the rate of cardiotoxicity of Doxil in patients treated with only about 100 mg/m2 total accumulated dose, the dose to be utilized here. The drug has been used in a few patients in the primary systemic therapy setting, with no reported clinical cardiotoxicity.

The expectation is that clinical and subclinical rates of cardiotoxicity will be very low or negligible at the total doses to be used here.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed, measurable, invasive breast carcinoma T >2cm, Nany, M0.
* Patients with node-negative, ER or PR-positive tumors ≤4 cm in size whose tumors are low risk (defined as a score of 0-17) on an Oncotype DX profile are not eligible.
* 19 years of age or greater
* Known ER, PR and HER-2 status (FISH assay to be done on specimens with 2+ or 3+ immunohistochemical staining for HER-2): patients with gene amplification on FISH study will be considered to be HER-2 positive. Patients for this study must be FISH negative if immunohistochemical stain is 2+ or 3+ positive; patients with negative, 0 or 1+ immunohistochemical stain for HER-2 are eligible.
* Known axillary nodal status: aspiration cytology or biopsy
* Documented menopausal status premenopausal (having menstrual periods or FSH <35) or postmenopausal (≥12 months since last menstrual period with intact uterus and at least one ovary or FSH ≥35 or previous bilateral oophorectomy
* Non-pregnant if premenopausal (negative serum or urine pregnancy test within 7 days of starting chemotherapy) and not breast feeding
* Patients with reproductive potential must use an adequate contraceptive method (e.g., abstinence, intrauterine device, barrier device with spermicide or surgical sterilization) during treatment and for three months after completing treatment.
* Life expectancy of less than 12 weeks
* Current, recent (within 4 weeks of the first infusion of this study), or planned participation in an experimental drug study other than a Genentech-sponsored Avastin cancer study
* Pregnant or lactating women.
* History of cardiac disease, with New York Heart Association Grade II or greater or clinical evidence of congestive heart failure.
* Serious comorbid medical conditions which would impair the ability to receive chemotherapy on time
* Previous invasive cancer within the last 5 years
* Altered mental status or dementia which would interfere with understanding of informed consent and ability to comply with study and follow-up procedures.
* Hypersensitivity to Doxil, doxorubicin, cyclophosphamide, cremophore (contained in teniposide, cyclosporine, and vitamin K), or to any component of Avastin
* Inadequately controlled hypertension (defined as blood pressure of >150/100 mmHg on antihypertensive medication)
* Unstable angina pectoris
* History of myocardial infarction or unstable angina within 12 months prior to beginning therapy
* History of stroke or TIA at any time
* Clinically significant vascular (e.g., aortic aneurysm requiring surgical repair or recent peripheral arterial thrombosis, aortic dissection) or peripheral vascular disease with 6 months prior to beginning therapy
* History of hemoptysis (greater than or equal to 1/2 teaspoon of bright red blood per episode) within 1 month prior to beginning therapy
* Evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation)
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to beginning therapy or anticipation of need for major surgical procedure during the course of the study
* Patients must have a 2-d echocardiogram indicating an ejection fraction of > 50% within 42 days prior to first dose of study drug. The method used at baseline must be used for later monitoring.
* No distant metastases on bone scan and on CT scans of chest and abdomen (no metastasis on optional PET scan is an acceptable alternative; if PET scan is done for any reason it must show no evidence of distant metastasis). Baseline PET scan is recommended but not required for all patients.
* No CNS metastasis
* Hbg ≥9 gm, platelets ≥100,000, granulocytes ≥1000, total or direct bilirubin ≤1.2, creatinine ≤2.0 and urine protein:creatinine ratio <1.0
* No prior chemotherapy or radiotherapy and ≤4 weeks of prior antiestrogen or aromatase inhibitor therapy
* No concomitant hormone replacement (i.e. estrogen or progestin) therapy
* PS less than or equal to one

Exclusion Criteria:

* Minor surgical procedure (excluding placement of a vascular access device) such as fine needle aspiration or core needle biopsy within 7 days of beginning therapy
* Urine protein:creatinine ratio ≥1.0 at initial screening
* Known hypersensitivity to any component of Avastin
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months of beginning therapy
* Serious, non-healing wound, active ulcer, or untreated bone fracture
* Any prior history of hypertensive crisis or hypertensive encephalopathy
* Known CNS metastasis, except for treated brain metastasis. Treated brain metastases are defined as having no evidence of progression or hemorrhage after treatment and no ongoing requirement for dexamethasone, as ascertained by clinical examination and brain imaging (MRI or CT) during the screening period. Anticonvulsants (stable dose) are allowed. Treatment for brain metastases may include whole brain radiotherapy (WBRT), radiosurgery (RS; Gamma Knife, LINAC, or equivalent) or a combination as deemed appropriate by the treating physician. Patients with CNS metastases treated by neurosurgical resection or brain biopsy performed within 3 months prior to Day 1 will be excluded.

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2008-03; Primary Completion 2014-12 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Carpenter, M.D., Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Doxil, Paclitaxel, Cyclophosphamide + Avastin: Two stage phase II single arm trial to evaluate the pathologic complete response rate to sequential dose dense chemotherapy using Doxil, paclitaxel and cyclophosphamide with concurrent Avastin in patients with locally advanced invasive breast cancer.
  Doxil, Paclitaxel, Cyclophosphamide, Avastin: Regimen A: Sequential Doxil 25 mg/m2 every 2 weeks for 3 doses, followed by paclitaxel 175 mg/m2 i.v. every 2 weeks for 3 doses, then cyclophosphamide 600 mg/M 2 i.v. every 2 weeks for 3 doses. Avastin 10 mg/kg i.v. every 2 weeks will be given concurrently with all 3 agents. Patients who experience <pCR to primary chemotherapy will receive an additional year of Avastin at the same dose equivalent beginning 6-8 weeks after definitive operation.
  Regimen B: Sequential Doxil 30 mg/m2 every 2 weeks for 3 doses will be followed by paclitaxel 175 mg/m2 i.v. every 2 weeks for 3 doses, then by cyclophosphamide 600 mg/m 2 i.v. every 2 weeks for 3 doses. Avastin 10 mg/kg i.v. every 2 week
Period: Overall Study
Arm/Group | Doxil, Paclitaxel, Cyclophosphamide + Avastin
Started | 32 (No patient received regimen B due to grade 3 toxicity in the third patient treated on regimen A.)
Completed | 31 (Followup through 10 years planned.)
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: women with locally advanced invasive breast cancer
Groups:
- Doxil, Paclitaxel, Cyclophosphamide + Avastin: Two stage phase II single arm trial to evaluate the pathologic complete response rate to sequential dose dense chemotherapy using Doxil, paclitaxel and cyclophosphamide with concurrent Avastin in patients with locally advanced invasive breast cancer.
  Regimen A: Sequential Doxil 25 mg/m2 every 2 weeks for 3 doses, then paclitaxel 175 mg/m2 i.v. every 2 weeks for 3 doses, then cyclophosphamide 600 mg/M 2 i.v. every 2 weeks for 3 doses. Avastin 10 mg/kg i.v. every 2 weeks will be given concurrently with all 3 agents. Patients who experience <pCR to chemotherapy will receive an additional year of Avastin at the same dose equivalent starting 6-8 weeks after operation.
  Regimen B: Identical to Regimen A except that the dose of Doxil will be 30 mg/m2.
Arm/Group | Doxil, Paclitaxel, Cyclophosphamide + Avastin
Number analyzed (Participants) | 32
Age, Continuous [Median (Full Range); unit: years] | 49 [34 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 32

OUTCOME MEASURES:

1. Primary Outcome: Rate of Achievement of Pathological Complete Response (pCR)
Description: Results of the pathologic evaluation of the surgical specimen(s) from operation (segmental or total mastectomy) will be used to report the overall complete pathological response rate. Criteria used were those described by Kaufmann et al, Journal of Clinical Oncology 2003; 21(13):2600-2608. The definition of pCR used from this source was absence of invasive cancer in both resected breast tissue and in resected axillary nodes.
Time Frame: After completion of at least 8 of the 9 chemotherapy doses and operation.
Population: Intention to treat, i.e., all participants entered were included in the analysis.
Measure: Number; unit: pathology specimens from participants
Groups:
- Doxil, Paclitaxel, Cyclophosphamide + Avastin: Two stage phase II single arm trial to evaluate the pathologic complete response rate to sequential dose dense chemotherapy using Doxil, paclitaxel and cyclophosphamide with concurrent Avastin in patients with advanced invasive breast cancer.
  Regimen A: Doxil 25 mg/M2 iv and Avastin 10 mg/kg iv every 2 weeks x 3, then paclitaxel 175 mg/M2 i.v. and Avastin 10 mg/kg iv every 2 weeks x 3, then cyclophosphamide 600 mg/M2 i.v. and Avastin 10 mg/kg iv every 2 weeks x 3 . Patients who experience <pCR to primary chemotherapy will receive an additional year of Avastin 15 mg/kg iv every 3 weeks, beginning 6-8 weeks after operation.
  Regimen B: Identical to Regimen A except that the Doxil dose was 30 mg/M2 iv every 2 weeks x 3.
Arm/Group | Doxil, Paclitaxel, Cyclophosphamide + Avastin
Number analyzed (Participants) | 32
pathology specimens from participants | 9
Statistical Analysis 1: Comparison: Doxil, Paclitaxel, Cyclophosphamide + Avastin; Test type: Superiority or Other; Hazard Ratio (HR) = 0.28

2. Secondary Outcome: Number of Participant With Clinical or Subclinical Cardiotoxicity
Description: Left ventricular ejection fraction (LVEF) measurements and clinical examination at baseline and at end of therapy will be used.
Time Frame: Prior to treatment and at completion of chemotherapy
Measure: Number; unit: participants
Groups:
- Doxil, Paclitaxel, Cyclophosphamide + Avastin: Two staged phase II single arm trial to evaluate the pathologic complete response rate to sequential dose dense chemotherapy using Doxil, paclitaxel and cyclophosphamide with concurrent Avastin in patients with advanced invasive breast cancer.
  Regimen A: Doxil 25 mg/M2 iv and Avastin 10 mg/kg iv every 2 weeks x 3, then paclitaxel 175 mg/M2 i.v. and Avastin 10 mg/kg iv every 2 weeks x 3, then cyclophosphamide 600 mg/M2 i.v. and Avastin 10 mg/kg iv every 2 weeks x 3 . Patients who experience <pCR to primary chemotherapy will receive an additional year of Avastin 15 mg/kg iv every 3 weeks, beginning 6-8 weeks after operation.
  Regimen B: Identical to Regimen A except that the Doxil dose was 30 mg/M2 iv every 2 weeks x 3.
Arm/Group | Doxil, Paclitaxel, Cyclophosphamide + Avastin
Number analyzed (Participants) | 31
participants | 0

3. Secondary Outcome: Calculate Progression Free Survival
Description: Progression free survival (PFS) will be defined as survival without local recurrence of breast cancer and without the development of distant metastasis. Death from any cause will be included as an event. The Kaplan-Meier nonparametric method will be used to estimate progression free survival.
Time Frame: 5 years
Population: operative specimens after treatment of participants
Measure: Number; unit: participants
Groups:
- Doxil, Paclitaxel, Cyclophosphamide + Avastin: Two stage phase II single arm trial to evaluate the pathologic complete response rate to sequential dose dense chemotherapy using Doxil, paclitaxel and cyclophosphamide with concurrent Avastin in patients with locally advanced invasive breast cancer.
  Doxil, Paclitaxel, Cyclophosphamide, Avastin:
  Regimen A: Doxil 25 mg/M2 iv and Avastin 10 mg/kg iv every 2 weeks x 3, then paclitaxel 175 mg/M2 i.v. and Avastin 10 mg/kg iv every 2 weeks x 3, then cyclophosphamide 600 mg/M2 i.v. and Avastin 10 mg/kg iv every 2 weeks x 3 . Patients who experience <pCR to primary chemotherapy will receive an additional year of Avastin 15 mg/kg iv every 3 weeks, beginning 6-8 weeks after operation.
  Regimen B: Identical to Regimen A except that the Doxil dose was 30 mg/M2 iv every 2 weeks x 3.
Arm/Group | Doxil, Paclitaxel, Cyclophosphamide + Avastin
Number analyzed (Participants) | 32
participants | 22

4. Secondary Outcome: Assess Toxicities of Regimen Including Hand Foot Syndrome
Description: patients who receive any treatment drugs will be included for toxicity evaluation. Adverse events will be summarized with frequencies and proportions of study participants exhibiting adverse events. The severity of adverse events (none, mild, moderate, severe) and their relationship to the product will be presented.
Time Frame: Baseline, every 2 weeks during treatment, and at completion of therapy. Every 3 weeks during postoperative Avastin
Measure: Number; unit: participants
Arm/Group | Doxil, Paclitaxel, Cyclophosphamide + Avastin
Number analyzed (Participants) | 32
participants | 23

ADVERSE EVENTS:
Time Frame: At baseline, every 2 weeks during chemotherapy and Avastin, every 3 weeks during postoperative Avastin, every 6 months afterward though 5 years of followup, then annually to 10 years of followup.
Groups:
- Doxil, Paclitaxel, Cyclophosphamide + Avastin: Two staged phase II single arm trial to evaluate the pathologic complete response rate to sequential dose dense chemotherapy using Doxil, paclitaxel and cyclophosphamide with concurrent Avastin in patients with advanced invasive breast cancer.
  Doxil, Paclitaxel, Cyclophosphamide, Avastin: Regimen A: Sequential Doxil 25 mg/m2 every 2 weeks for 3 doses will be followed by paclitaxel 175 mg/m2 i.v. every 2 weeks for 3 doses, then by cyclophosphamide 600 mg/M 2 i.v. every 2 weeks for 3 doses. Avastin 10 mg/kg i.v. every 2 weeks will be given concurrently with all 3 agents. Patients who experience <pCR to primary chemotherapy will receive an additional year of Avastin at the same dose equivalent beginning 6-8 weeks after definitive operation.
  Regimen B: Sequential Doxil 30 mg/m2 every 2 weeks for 3 doses will be followed by paclitaxel 175 mg/m2 i.v. every 2 weeks for 3 doses, then by cyclophosphamide 600 mg/m 2 i.v. every 2 weeks for 3 doses. Avastin 10 mg/kg i.v. every 2 week
Arm/Group | Doxil, Paclitaxel, Cyclophosphamide + Avastin
Serious Adverse Events (participants affected / at risk) | 1/32
Other Adverse Events (participants affected / at risk) | 23/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Doxil, Paclitaxel, Cyclophosphamide + Avastin (N=32)
hospitalization (Skin and subcutaneous tissue disorders) | 1 (1) — Transferred to hospital from an outside institution because of suspected Stevens-Johnson syndrome. Found to have grade 3 hand-foot syndrome. Sent home on 3rd day after symptomatic treatment, then she resumed and completed her preoperative treatment.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Doxil, Paclitaxel, Cyclophosphamide + Avastin (N=32)
rash (Skin and subcutaneous tissue disorders) | 17 (17) — any grade
hand-foot syndrome (Skin and subcutaneous tissue disorders) | 23 (23) — palmar-plantar erythrodysesthesia, any grade. 1 participant had grade 3 event
mucositis (Gastrointestinal disorders) | 1 (1) — grade 3
proteinuria (Renal and urinary disorders) | 1 (1) — grade 3
hypertension (General disorders) | 7 (7) — grade 3
neutropenia (Blood and lymphatic system disorders) | 6 (6) — grade 3

LIMITATIONS AND CAVEATS:
pilot study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No